CLINICAL TRIAL: NCT07198919
Title: Comparison of Inter-appointment Pain Reduction During Root Canal Treatment in Symptomatic Apical Periodontitis by Using Intracanal Medicaments Chlorhexidine Gel and Single Antibiotic Paste Nitrofurantoin
Brief Title: Comparison of Inter-appointment Pain Reduction During Root Canal Treatment in Symptomatic Apical Periodontitis by Using Intracanal Medicaments; Chlorhexidine Gel and Single Antibiotic Paste Nitrofurantoin
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Altamash Institute of Dental Medicine (Other)
Responsible Party: Principal Investigator, Fiza Bibi Alavi, FCPS II Resident Trainee, Altamash Institute of Dental Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIDM/ERC/03/2025/01
Record Dates: First submitted 2025-05-28; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-05

CONDITIONS: Intracanal Medicament
Keywords: intracanal medicament
MeSH Terms: interventions — Nitrofurantoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Chlorhexidine (Active Comparator)
  Interventions: Drug: Chlorhexidine gel
- Nitrofurantoin (Active Comparator)
  Interventions: Drug: Nitrofurantoin 100 MG

INTERVENTIONS:
Drug: Chlorhexidine gel — 0.12% Chlorhexidine gel (Consepsis Ultradent)
  Other Names: Consepsis Ultradent
  Arms: Chlorhexidine
Drug: Nitrofurantoin 100 MG — Nitrofurantoin Tablets 100mg
  Arms: Nitrofurantoin

SUMMARY:
This study is being conducted to find out which of two medications-Chlorhexidine Gel or Nitrofurantoin-works better in reducing pain between root canal treatment visits. Sometimes, patients with infected teeth (called symptomatic apical periodontitis) continue to feel pain between treatment appointments. To help with this, dentists use medications inside the cleaned tooth canal.

In this trial, 220 patients will be divided into two groups. One group will receive Chlorhexidine Gel, and the other will receive Nitrofurantoin paste inside their tooth during the first treatment visit. Pain levels will be recorded before treatment, and again after 24 and 48 hours using a pain scale from 0 (no pain) to 10 (severe pain). No pain medicine will be given unless the patient feels very uncomfortable.

The study is taking place at the Altamash Institute of Dental Medicine in Karachi, and will help dentists understand which medication helps patients feel better faster during root canal treatment.

DETAILED DESCRIPTION:
This randomized controlled trial is designed to evaluate and compare the efficacy of two commonly used intracanal medicaments-2% Chlorhexidine Gel and Single Antibiotic Paste (Nitrofurantoin)-in reducing inter-appointment pain during root canal treatment of teeth diagnosed with symptomatic apical periodontitis.

Pain between root canal visits is a common concern. The persistence of microbial infection within the root canal system can lead to inflammation of the peri-radicular tissues, causing discomfort. Intracanal medicaments are placed after chemo-mechanical preparation to enhance disinfection, reduce microbial load, and minimize postoperative complications such as pain.

While Chlorhexidine has long been used due to its broad-spectrum antimicrobial activity and substantivity, Nitrofurantoin, a nitrofuran antibiotic, has shown promising results against resistant organisms and may offer similar or enhanced pain relief when used as a local medicament.

A total of 220 patients, aged 16 to 45 years, presenting with single-rooted permanent teeth requiring primary root canal treatment and diagnosed with pulp necrosis and symptomatic apical periodontitis, will be enrolled at the Department of Operative Dentistry and Endodontics, Altamash Institute of Dental Medicine, Karachi. Patients will be randomly allocated into two equal groups (n=110 per group) using the lottery method.

Group 1 will receive Chlorhexidine Gel as the intracanal medicament.

Group 2 will receive Nitrofurantoin Paste, prepared by mixing crushed Nitrofurantoin tablets with saline.

Pain intensity will be measured using the Visual Analogue Scale (VAS) at three time points: preoperatively, 24 hours, and 48 hours after the first treatment visit. Inter-appointment pain reduction will be calculated using the formula:

[(Pre-treatment VAS score - Post-treatment VAS score) / Pre-treatment VAS score] × 100

Standardized root canal procedures, including anesthesia, canal preparation, irrigation, medicament placement, and obturation, will be performed by a single postgraduate trainee to ensure consistency. No analgesics will be prescribed unless requested by the patient due to severe discomfort. If needed, ibuprofen 200 mg will be provided and documented.

Data will be analyzed using SPSS version 20. Continuous variables (e.g., pain scores) will be assessed for normality. Depending on distribution, t-tests or non-parametric equivalents will be used to compare groups. Stratification will be done for potential confounders such as age, gender, and type of tooth. A p-value < 0.05 will be considered statistically significant.

The study's goal is to provide evidence on whether Nitrofurantoin is more effective than Chlorhexidine Gel in reducing pain between appointments, potentially offering a new and effective intracanal medicament option in endodontic practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with single rooted permanent teeth of both arches.
* Patients with a pulpal status of necrosis with or without periapical radiolucency, confirmed using Electric Pulp Test (EPT) and Cold Test.
* Male and female patients age of 16 to 45 yrs.
* Patients of both genders.

Exclusion Criteria:

* Patients with uncontrolled diabetes.
* Presence of periapical granuloma or cyst confirmed via radiographic evaluation.
* Patient is on any medication that affects pain, inflammation and infection like analgesic, antibiotics since last 7 days
* Patient requiring endodontic re-treatment.
* Patients with immature teeth with open apices.
* Patients with calcified canals.

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Percentage Reduction in Inter-Appointment Pain Score | Pain scores will be assessed before treatment, then at 24 hours and 48 hours after the first treatment visit.
  Change in patient-reported pain intensity, measured using the Visual Analogue Scale (VAS), from pre-treatment to 24 and 48 hours post-treatment. Pain reduction will be calculated using the formula:
  [(Pre-treatment VAS score - Post-treatment VAS score) / Pre-treatment VAS score] × 100

CONTACTS AND LOCATIONS:
Locations (1):
- AIDM, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided